CLINICAL TRIAL: NCT02916329
Title: Targeted Molecular Imaging of [68Ga]- Labelling Anti-EGFR Affibody Molecule in EGFR ECD in Lung Cancer Patients and Healthy Volunteers
Brief Title: In Vivo EGFR-ECD Molecular Imaging Using [68Ga]- Labelling Anti-EGFR Affibody Molecule
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Xilin Sun, Chief, Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 14402
Record Dates: First submitted 2016-09-24; First posted 2016-09-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Molecular Imaging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 68Ga-ZEGFR: EGFR++ (Experimental): Patients in this group had EGFR-activating mutant and EGFR high expression tumors and did not receive any treatment before this study.
  Interventions: Other: 68Ga-NODAGA-Ac-Cys-ZEGFR:1907
- 68Ga-ZEGFR: EGFR+ (Experimental): Patients in this group had EGFR-activating mutant and EGFR medium expression tumors and did not receive any treatment before this study.
  Interventions: Other: 68Ga-NODAGA-Ac-Cys-ZEGFR:1907
- 68Ga-ZEGFR: EGFR- (Experimental): Patients in this group had no EGFR expression tumors and did not receive any treatment before this study.
  Interventions: Other: 68Ga-NODAGA-Ac-Cys-ZEGFR:1907
- 68Ga-ZEGFR: EGFR wild type (Experimental): Patients in this group had EGFR wild-type tumors and did not receive any treatment before this study.
  Interventions: Other: 68Ga-NODAGA-Ac-Cys-ZEGFR:1907
- 68Ga-ZEGFR:unknown EGFR status (Experimental): Patients without the EGFR status measurement results and did not receive any treatments were classified in this group.
  Interventions: Other: 68Ga-NODAGA-Ac-Cys-ZEGFR:1907
- 68Ga-ZEGFR: EGFR (Experimental): Patients in this group had EGFR expression tumors and had receive some treatment before this study.
  Interventions: Other: 68Ga-NODAGA-Ac-Cys-ZEGFR:1907

INTERVENTIONS:
Other: 68Ga-NODAGA-Ac-Cys-ZEGFR:1907 — 68Ga-NODAGA-Ac-Cys-ZEGFR:1907 (Ac-Cys-ZEGFR:1907 : Ac-CVDNKFNKEMWAAWE EIRNLPNLN GWQMTAFIASLVDDPSQSANLLAEAKKLNDAQAPK-NH2)

SUMMARY:
The investigators developed [68Ga]-labelling Anti-EGFR Affibody Molecule as a targeted molecular imaging agent for noninvasive and repeatable detecting EGFR-ECD expression status.

DETAILED DESCRIPTION:
The goals of investigators are to evaluate the use of [68Ga]-labelling Anti-EGFR Affibody Molecule as a novel PET/CT radiotracer to monitor EGFR-ECD expression status and classify EGFR-ECD benefit NSCLC patients. The investigators want to evaluated the use of [68Ga]-labelling Anti-EGFR Affibody Molecule in lung cancer imaging in adult NSCLC patients with different EGFR-ECD expression status of primary and metastatic cancers.

ELIGIBILITY:
Inclusion Criteria:

* Advanced NSCLC
* 18 years or older
* A life expectancy of at least 12 weeks
* Presence of a malignant lesion within the chest of at least 0.5 cm diameter as measured by computed tomography (CT)
* Written informed consent

Exclusion Criteria:

* Claustrophobia
* Pregnancy
* Metal implants in the thorax

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-09; Primary Completion 2016-10 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
tumor SUVmax value of 68Ga-NODAGA-ZEGFR:1907 PET/CT Imaging | at time of imaging
  To quantify the accumulation, a volume of interest using a 3-D sphere, was placed over the primary lung tumor, lymph nodes and distant metastases avoiding necrosis, blood vessels and normal lung tissue as much as possible on a workstation (Advantage Workstation 4.6; GE Healthcare). The maximum standard uptake value (SUVmax) normalized to body weight (kBq/mL) was calculated within the region of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Shen Baozhong, M.D., Study Chair — The Fourth Hospital of Harbin Medical University
Locations (1):
- TOF-PET/CT/MR center of the Fourth Hospital of Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: Undecided